CLINICAL TRIAL: NCT02582424
Title: Safety and Efficacy of PDL-0101 in Patients With Hyperlipidemias: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDT-0101
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-10

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDL-0101 (Experimental): EPA +astaxanthin
  Interventions: Other: PD-L0101
- placebo (Placebo Comparator): olive oil
  Interventions: Other: placebo

INTERVENTIONS:
Other: PD-L0101 — 92% EPA+6 mg ATX+50 mg TCT GG BID
  Arms: PDL-0101
Other: placebo — placebo
  Arms: placebo

SUMMARY:
This will be an 8 week multicenter, randomized, double-blind, placebo controlled trial.

DETAILED DESCRIPTION:
This will be an 8 week, multicenter, randomized, double blind, placebo controlled trial. The screening visit will be divided into two parts, a "pre-screen" in-clinic rapid lipid test (Cholestech) followed by a full screening blood draw to be sent to the central reference laboratory (CRL) for subjects meeting the Cholestech inclusion values for TG and LDL (see inclusion criteria below) on the pre-screen test. Subjects who do not meet the pre-screen criteria will be discharged from further participation in the study. Subjects must have pre-screen lipid values of LDL >/=70 mg/dl and triglyceride (TG) >/=180 and </=499. Subjects who meet these Cholestech criteria will have blood drawn for central reference laboratory (CRL) screening testing. For randomization, 80% of the subjects must have TG>/=200 mg/dl to proceed to the next screening step while up to 20% will be allowed to proceed to the next screening step with TG=150-199 mg/dl as long as the LDL is>/=70 mg/dl. Subjects who meet the CRL pre-screen lipid inclusion criteria will return 2-14 days later for the remainder of the full screening procedures. Subjects who meet all screening criteria will be randomized at this visit. Thus, the prescreening and screening-1 visits will occur at the same time and the screening 2 visit will also be the baseline visit. BMI will be calculated but is not a criterion for participation.

Subjects who meet all inclusion and exclusion requirements at the screening 2/baseline visit will be randomized to receive one of the two (2) study products. Randomization will proceed in groups of 5 with 4 subjects having TG between 200-499 mg/dl before randomizing a subject with TG between 150-199 mg/dl. Subjects will return for evaluation 4 and 8 weeks after the baseline visit at which times adverse events (AEs) will be recorded, blood lipid studies will be done and subjects will complete a VAS for product tolerability. Laboratory studies will be drawn after subjects have been sitting for at least 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Either gender, in general good health, between 25-85 years old
2. Serum TG 150-495 mg/dl at screening
3. Serum LDL >/= 70 mg/dl at screening
4. Not using any other product including drugs, medical foods, neutraceuticals or dietary supplements for control of serum lipids
5. Consistent dietary habits
6. Women of child bearing potential must use an accepted method of birth control
7. Able to read and understand study documents including the Subject Informed Consent Document (Spanish language translation available, if needed)

Exclusion Criteria:

1. serum TG <150 or >495 mg/dl at screening visit
2. serum LDL<50 mg/dl at screening visit
3. use of any other serum lipid modifying agent (see section 6.0) within 4 weeks of screening visit
4. history of any intestinal disease that might interfere with absorption
5. history of pancreatitis, inflammatory colitis or prior cholecystectomy
6. any active malignancy or history of malignancy, except basal cell carcinoma or cervical carcinoma in situ curatively treated, within 3 years of the screening visit
7. screening AST, ALT, alkaline phosphatase, bilirubin >1.3 times the upper limit of normal for the reference laboratory
8. serum creatinine >2.0
9. uncontrolled diabetes mellitus (glycosylated Hgb >9)
10. diabetes mellitus not on stable therapy for at least 2 months
11. uncontrolled hypertension (DBP >100, SPB >160)
12. unstable angina, congestive heart failure or other uncontrolled cardiac disease
13. pregnant or lactating women
14. known history of allergies to O-3 fatty acids, carotenoids, vitamin E or fish products
15. history of substance abuse or any psychiatric condition that may impair the subject's ability to comply with the study requirements.
16. Regular consumption of more than one (1) unit of alcohol daily. For the purposes of this study a unit of alcohol consists of 12 oz. of beer, 6 oz. of wine or 2 oz of hard spirits.
17. any medical condition that, in the opinion of the investigator, might put the subject at undue risk or might interfere with the subject's ability to participate in the study
18. participation in another clinical trial within 30 days or 6 half lives of the study agent, whichever is longer, of the screening visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
lowering serum TG levels | 8 weeks
  more effective than placebo at lowering serum TG levels

SECONDARY OUTCOMES:
lower serum LDL levels | 8 weeks
  lower serum LDL levels

CONTACTS AND LOCATIONS:
Overall Officials: Jay Udani, MD, Principal Investigator — Medicus Research 18250 Roscoe Blvd. Northridge CA 91325; Andrea Lawless, MD, Principal Investigator — Provident Clinical Research 211 E Lake St. Addison IL 60101